CLINICAL TRIAL: NCT01263106
Title: Effect of LY2216684 on the Pharmacokinetics of Theophylline in Healthy Subjects
Brief Title: A Study of LY2216684 and Theophylline in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 12594; H9P-EW-LNCE (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-12-16; First posted 2010-12-20 (Estimated); Results first posted 2019-07-08 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-04

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — alpha-((5-fluoro-2-methoxyphenyl)methyl)-alpha-(tetrahydro-2H-pyran-4-yl)-2-morpholinemethanol; Theophylline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Theophylline, LY2216684 + Theophylline (Experimental): Period 1: single 200-milligram (mg) theophylline oral dose on Day 1; Washout period of at least 7 days; Period 2: 18 mg LY2216684 orally, once daily on Days 1-5 with single 200-mg theophylline oral dose coadministered on Day 3
  Interventions: Drug: LY2216684; Drug: Theophylline
- LY2216684 + Theophylline, Theophylline (Experimental): Period 1: 18 mg LY2216684 orally, once daily on Days 1-5 with single 200-mg theophylline oral dose coadministered on Day 3; Washout period of at least 7 days; Period 2: single 200-mg theophylline oral dose on Day 1
  Interventions: Drug: LY2216684; Drug: Theophylline

INTERVENTIONS:
Drug: LY2216684 — 18-mg LY2216684 oral dose
Drug: Theophylline — 200-mg theophylline oral dose

SUMMARY:
The primary objective of this study is to confirm that LY2216684 is not an inhibitor of cytochrome P450 1A2 (CYP1A2) in healthy participants using theophylline as a probe substrate for the enzyme. Because LY2216684 has been observed to increase heart rate in some healthy participants, this study will also assess heart rate when coadministered with theophylline.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy males or females, as determined by medical history and physical examination.
* Male participants - Agree to use a reliable method of birth control during the study and for 1 month following the last dose of study drug.
* Female participants - Are women of child-bearing potential who test negative for pregnancy at the time of enrollment, have used a reliable method of birth control for 6 weeks prior to administration of study drug and agree to use a reliable method of birth control both during the study and for 1 month following the last dose of study drug; or are women not of child-bearing potential due to surgical sterilization (hysterectomy or bilateral oophorectomy or tubal ligation) or menopause (at least 1 year without menses or 6 months without menses and a follicle stimulating hormone [FSH] >40 mass International Units per milliliter [mIU/mL]).
* Have body weight >50 kilograms (kg).
* Have clinical laboratory test results within normal reference range for the population or investigator site, or results with acceptable deviations that are judged to be not clinically significant by the investigator.
* Have venous access sufficient to allow blood sampling as per the protocol.
* Have normal sitting blood pressure and pulse rate as determined by the investigator.
* Are reliable and willing to be available for the duration of the study and are willing to follow study procedures.
* Have given written informed consent approved by Lilly and the ethical review board (ERB) governing the site.

Exclusion Criteria:

* Are investigator site personnel directly affiliated with this study and their immediate families. Immediate family is defined as a spouse, parent, child or sibling, whether biological or legally adopted.
* Are currently enrolled in, or discontinued within the last 30 days from, a clinical trial involving an investigational drug or device or off-label use of a drug or device other than the study drug, or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study.
* Have known allergies to LY2216684, theophylline, or related compounds.
* Are persons who have previously completed or withdrawn from this study or any other study investigating LY2216684 within 6 months prior to screening.
* Have an abnormality in the 12-lead electrocardiogram (ECG) that, in the opinion of the investigator, increases the risks associated with participating in the study.
* Have a history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data.
* Have a history or show evidence of significant active neuropsychiatric disease or have a history of suicide attempt or ideation.
* Regularly use known drugs of abuse and/or show positive findings on urinary drug screening.
* Show evidence of human immunodeficiency virus (HIV) and/or positive human HIV antibodies.
* Show evidence of hepatitis C and/or positive hepatitis C antibody.
* Show evidence of hepatitis B and/or positive hepatitis B surface antigen.
* Are women with a positive pregnancy test or women who are lactating.
* Intend to use over-the-counter or prescription medication within 14 days prior to dosing unless deemed acceptable by the investigator and Sponsor's medical monitor.
* Use of any drugs or substances that are known to be substrates, inducers, or inhibitors of cytochrome P450 1A2 (CYP1A2) within 30 days prior to dosing.
* Have donated blood of more than 500 mL within the last month.
* Have an average weekly alcohol intake that exceeds 14 units per week, or are unwilling to stop alcohol consumption for 48 hours prior to check-in in each period and while resident at the clinical research unit (CRU) (1 unit = 12 ounces [oz] or 360 mL of beer; 5 oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits).
* Consume 5 or more cups of coffee (or other beverages of comparable caffeine content) per day, on a habitual basis, or any participants unwilling to adhere to study caffeine and chocolate restrictions.
* Have used any tobacco-containing or nicotine-containing products (including but not limited to cigarettes, pipes, cigars, chewing tobacco, nicotine patches, nicotine lozenges, or nicotine gum) within 6 months prior to enrollment.
* Have consumed grapefruit or grapefruit-containing products 7 days prior to enrollment and during the study.
* Have a documented or suspected history of glaucoma.
* Participants determined to be unsuitable by the investigator for any reason.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2010-12; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Theophylline Alone, Then LY2216684 + Theophylline: Period 1: single 200 mg theophylline oral dose on Day 1; Washout period of at least 7 days; Period 2: 18 mg LY2216684 orally once daily on Days 1-5. Single dose of 200 mg theophylline coadministered on Day 3.
- LY2216684 + Theophylline, Then Theophylline Alone: Period 1: 18 mg LY2216684 orally once daily on Days 1-5. Single dose of 200 mg theophylline coadministered on Day 3.Washout period of at least 7 days; Period 2: single 200 mg theophylline oral dose on Day 1
Period: Period 1 (7 Days)
Arm/Group | Theophylline Alone, Then LY2216684 + Theophylline | LY2216684 + Theophylline, Then Theophylline Alone
Started | 11 | 10
Completed | 11 (Period 1: 1 participant took theophylline alone but was not given LY + theophylline.) | 10 (Period 1: 1 participant took LY + theophylline but was not given theophylline alone.)
Not Completed | 0 | 0
Period: Washout (at Least 7 Days)
Arm/Group | Theophylline Alone, Then LY2216684 + Theophylline | LY2216684 + Theophylline, Then Theophylline Alone
Started | 11 | 10
Completed | 10 | 9
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1
Period: Period 2 (7 Days)
Arm/Group | Theophylline Alone, Then LY2216684 + Theophylline | LY2216684 + Theophylline, Then Theophylline Alone
Started | 10 | 9
Completed | 10 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All started participants.
Arm/Group | All Participants
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.2 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics: Area Under the Plasma Concentration-Time Curve From Time 0 Hour to Infinity (AUC0-∞) of Theophylline
Description: The Least Squares (LS) geometric mean was based on AUC0-∞. The AUC for theophylline was calculated on Day 1 of a given period when theophylline was administered alone and on Day 3 of another period when theophylline was coadministered with LY2216684.
Time Frame: Predose 1, 2, 3, 4, 6, 8, 12, 24, 48, and 72 hours post-administration of theophylline on Days 1 and 3
Population: The safety population included participants who were randomized, received study drug, and had at least 1 post-dose safety assessment.
Measure: Geometric Mean (90% Confidence Interval); unit: nanogram*hour per milliliter (ng*h/mL)
Groups:
- Theophylline Alone: Single 200 mg theophylline oral dose on Day 1.
- LY2216684 + Theophylline: Oral dose of 18 mg LY2216684, once daily on Days 1-5 with single 200 mg theophylline dose coadministered on Day 3.
Arm/Group | Theophylline Alone | LY2216684 + Theophylline
Number analyzed (Participants) | 20 | 20
nanogram*hour per milliliter (ng*h/mL) | 70200 [62300 to 79200] | 78700 [69800 to 88800]
Statistical Analysis 1: Comparison: Theophylline Alone vs LY2216684 + Theophylline; Test type: Superiority or Other; Mixed Models Analysis; Ratio of Geometric LS Means = 1.12, 90% CI 2-sided [1.05 to 1.20]

2. Primary Outcome: Pharmacokinetics: Maximum Plasma Concentration (Cmax) of Theophylline
Description: The Least Squares (LS) geometric mean was based on Cmax for theophylline on Day 1 of a given period when theophylline was administered alone and on Day 3 of another period when theophylline was coadministered with LY2216684.
Time Frame: Predose 1, 2, 3, 4, 6, 8, 12, 24, 48, and 72 hours post-administration of theophylline on Days 1 and 3
Population: as for outcome 1
Measure: Geometric Mean (90% Confidence Interval); unit: nanogram per milliliter (ng/mL)
Groups:
- Theophylline: Single 200 mg theophylline oral dose on Day 1.
Arm/Group | Theophylline | LY2216684 + Theophylline
Number analyzed (Participants) | 20 | 20
nanogram per milliliter (ng/mL) | 3174.35 [2796.84 to 3602.81] | 3054.84 [2691.79 to 3466.97]
Statistical Analysis 1: Comparison: Theophylline vs LY2216684 + Theophylline; Test type: Superiority or Other; Mixed Models Analysis; Ratio of Geometric LS Means = 0.96, 90% CI 2-sided [0.92 to 1.01]

3. Primary Outcome: Pharmacokinetics: Time to Maximum Plasma Concentration (Tmax) of Theophylline
Description: This outcome was measured based on Tmax for theophylline on Day 1 of a given period when theophylline was administered alone and on Day 3 of another period when theophylline was coadministered with LY2216684.
Time Frame: Predose 1, 2, 3, 4, 6, 8, 12, 24, 48, and 72 hours post-administration of theophylline on Days 1 and 3
Population: as for outcome 1
Measure: Median (Full Range); unit: hour (h)
Arm/Group | Theophylline | LY2216684 + Theophylline
Number analyzed (Participants) | 19 | 19
hour (h) | 12.00 [4.00 to 12.03] | 12.00 [3.00 to 12.00]
Statistical Analysis 1: Comparison: Theophylline vs LY2216684 + Theophylline; Test type: Superiority or Other; p = 0.8008, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.00, 90% CI 2-sided [-3.00 to 1.00]

4. Secondary Outcome: Mean Change From Baseline in Heart Rate: 200 mg Theophylline
Time Frame: Baseline, Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Theophylline
Number analyzed (Participants) | 20
beats per minute (bpm)
  Day 1 (-2 to 0 hours) | 74.1 (8.9)
  Day 1 (23 to 24 hours) | 82.7 (9.5)

5. Secondary Outcome: Mean Change From Baseline in Heart Rate: 18 mg LY221684 + 200 mg Theophylline
Time Frame: Baseline, Day 1, Day 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Groups:
- 18 mg LY2216684 + 200 mg Theophylline: Oral dose of 18 mg LY2216684, once daily on Days 1-5 with single 200 mg theophylline dose coadministered on Day 3.
Arm/Group | 18 mg LY2216684 + 200 mg Theophylline
Number analyzed (Participants) | 20
beats per minute (bpm)
  Day 1 (-2 to 0 hr) | 70.1 (7.2)
  Day 1 (23 to 24 hr): number analyzed (Participants) | 19
  Day 1 (23 to 24 hr) | 89.6 (9.1)
  Day 3 (-2 to 0 hr) | 74.1 (8.9)
  Day 3 (23 to 24 hr) | 95.7 (10.7)

ADVERSE EVENTS:
Description: During Period 1: 1 participant took theophylline alone but was not given LY + theophylline and 1 participant took LY + theophylline but was not given theophylline alone.
Groups:
- LY2216684: 18 mg LY2216684 orally
- Theophylline: single 200-mg theophylline oral dose
- LY2216684 + Theophylline: 18 mg LY2216684 orally with single 200-mg theophylline oral dose coadministered
Arm/Group | LY2216684 | Theophylline | LY2216684 + Theophylline
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 4/20 | 6/20 | 7/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2216684 (N=20) | Theophylline (N=20) | LY2216684 + Theophylline (N=20)
Palpitations (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 1 (1)
Feeling jittery (General disorders) | 1 (1) | 0 (0) | 1 (1)
Thirst (General disorders) | 0 (0) | 0 (0) | 1 (1)
Vessel puncture site pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days